CLINICAL TRIAL: NCT02355106
Title: A Prospective, Multicenter, Investigation of the Adagio PolarStar System in Subjects With Atrial Flutter
Brief Title: Prospective, Multicenter, Investigation of the Adagio Cryoablation System in Subjects With Atrial Flutter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adagio Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-001
Record Dates: First submitted 2015-01-27; First posted 2015-02-04 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2017-12

CONDITIONS: Atrial Flutter
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Atrial flutter Ablation
  Interventions: Device: PolarStart System

INTERVENTIONS:
Device: PolarStart System — Atrial flutter Ablation

SUMMARY:
The objective of the study is to demonstrate the safety and feasibility of the Adagio System in subjects with Atrial Flutter.

ELIGIBILITY:
Inclusion Criteria:

* Two symptomatic episodes of typical AFl (or chronic atrial flutter) during the one-year period prior to enrollment. This may include typical AFl occurring while receiving anti-arrhythmic drug (AAD) therapy for non-AFl tachyarrhythmia, including atrial fibrillation (AF).
* At least one episode of typical (clockwise or counterclockwise) atrial flutter documented by 12 lead electrocardiogram (ECG) within 6 months prior to enrollment.
* Subject has been diagnosed with symptomatic AFl
* Subject is at least 18 and ≤75 years of age.
* Subject is able and willing to give informed consent

Exclusion Criteria:

* Intra-cardiac thrombus has not been eliminated in subjects exposed to less than 4 weeks of therapeutic anticoagulation and a TEE (trans-esophageal echocardiogram) and/or CT did not conclusively rule out thrombus
* Subject developed persistent AF at least once in history (electrical or pharmacological cardioversion after 48h or episode duration >7 days).

Subject had any previous left atrial ablation.

* Subject had any previous cardiac surgery, e.g. prosthetic valves, except in the case of an isolated coronary bypass surgery performed more than three months prior to the procedure.
* Subject has permanent pacemaker or defibrillator implant.
* Subject has 2° type II, 3° degree atrioventricular (AV) block or left/right bundle branch block pattern
* Subject has unstable angina pectoris.
* Subject has history of previous myocardial infarction (MI) or percutaneous intervention during the last three months or planned in the next 3 months.

Subject has symptomatic carotid stenosis.

* Subject has chronic obstructive pulmonary disease with detected pulmonary hypertension or any other evidence of significant lung disease.
* Subject has any contraindication for oral anticoagulation.
* Subject has any history of previous transient ischemic attack (TIA) or stroke.
* Subject has known intra-cardiac thrombus formation.
* Subject has any significant congenital heart defect corrected or not (except for patent foramen ovale that is allowed).
* Subject has evidence of congestive heart failure (NYHA class II, III or IV) in sinus rhythm.
* Subject has hypertrophic cardiomyopathy.
* Subject has abnormal long or short QT interval, signs of Brugada syndrome, known inheriting ion channel disease on the family, arrhythmogenic right ventricular dysplasia.
* Subject has sarcoidosis.
* Subject has myxoma.
* Subject has thrombocytosis (platelet count > 600,000 / μl) or thrombocytopenia (platelet count <100,000 / μl).
* Subject has any untreated or uncontrolled hyperthyroidism or hypothyroidism.
* Subject has renal dysfunction with glomerular filtration rate < 60 ml/min/1.72m2.
* Subject has a reversible causes for AF like alcoholism.
* Subject is a pregnant woman or woman of childbearing potential not on adequate birth control: only woman with a highly effective method of contraception [oral contraception or intra-uterine device] (who must have a negative pregnancy test within 1 week of randomization) or sterile woman can be enrolled.
* Subject is a breastfeeding woman.
* Subject has an active systemic infection.
* Subject is unwilling or unable to comply fully with study procedures and follow-up due to any disease condition, which can raise doubt about compliance and influencing the study outcome especially any kind of cancer requiring ongoing in-hospital treatment, severe bleeding in history or a suspected pro-coagulant state.
* Legal incapacity or evidence that a subject cannot understand the purpose and risks of the study or inability to comply fully with study procedures and follow up.
* Subject has a life expectancy of ≤ 1 year.
* Subject is participating in any other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-01; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Safety measured by the percentage of subjects experiencing cardiovascular specific adverse events (CSAE) within thirty 30 days of the ablation procedure. | 30 DAYS

SECONDARY OUTCOMES:
Acute Success measured by Percentage of subjects with termination of AFl and complete bidirectional conduction block across the subeustachian (cavo-tricuspid) isthmus at the end of the ablation procedure. | 30 minutes
Outcome success | 30 days
  Percent of subjects with absence of AFl at 30 days (30 day ECG and as reported by subject or holter monitor)

CONTACTS AND LOCATIONS:
Locations (2):
- OLV Hospital, Aalst, Belgium
- St. Antonius Hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] Klaver MN, De Potter TJR, Iliodromitis K, Babkin A, Cabrita D, Fabbricatore D, Boersma LVA. Ultralow temperature cryoablation using near-critical nitrogen for cavotricuspid isthmus-ablation, first-in-human results. J Cardiovasc Electrophysiol. 2021 Aug;32(8):2025-2032. doi: 10.1111/jce.15142. Epub 2021 Jul 9. PMID 34196991